CLINICAL TRIAL: NCT00463762
Title: Cefoperazone/Sulbactam In The Treatment Of Serious Intra-Abdominal And Hepatobiliary Infections In Slovakia. An Open, Prospective, Non-Comparative Study.
Brief Title: Cefoperazone/Sulbactam In The Treatment Of Serious Intra-Abdominal And Hepatobiliary Infections.
Status: Withdrawn | Type: Observational
Sponsor: Pfizer (Industry)
Other Study IDs: A1891004
Record Dates: First submitted 2007-04-17; First posted 2007-04-20 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Abscess, Intra-Abdominal; Cholecystitis; Wound Infections; Peritonitis; Appendicitis
MeSH Terms: conditions — Abdominal Abscess; Cholecystitis; Wound Infection; Peritonitis; Appendicitis | interventions — Sulbactam

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: CP-75385-02 Cefoperazone/sulbactam

SUMMARY:
The primary objective is to collect data on treatment outcomes (clinical and microbiological cure), safety and tolerability of treatment with cefoperazone/sulbactam in patients with serious intra-abdominal and hepatobiliary infections in Slovakia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of age 18 years or older.
* Patient with intraabdominal/hepatobiliary infection.?

Exclusion Criteria:

* Patients with known hypersensitivity to penicillins, cephalosporins, cefoperazone or to sulbactam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1891004&StudyName=Cefoperazone/Sulbactam%20In%20The%20Treatment%20Of%20Serious%20Intra-Abdominal%20And%20Hepatobiliary%20Infections.